CLINICAL TRIAL: NCT07284095
Title: SANTE INITIATIVE: Nutritional Intervention With Tenebrio Molitor Powder in Children With Chronic Malnutrition in the Democratic Republic of the Congo
Brief Title: Nutritional Intervention With Tenebrio Molitor Powder in Children With Chronic Malnutrition in the Democratic Republic of the Congo
Acronym: SANTE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: Fundación Amigos de Monkole (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SANTE
Record Dates: First submitted 2025-11-17; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Malnutrition; Stunting of Growth
Keywords: Chronic Malnutrition; Stunting; Tenebrio Molitor; Food Security; Sustainable Foods
MeSH Terms: conditions — Growth Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will receive a daily supplement made from Tenebrio molitor (mealworm) flour for 24 weeks.
  Interventions: Dietary Supplement: Tenebrio Molitor powder
- Control Group (Active Comparator): Participants will receive a daily supplement made from maize and soy flour for 24 weeks.
  Interventions: Dietary Supplement: Control Group (Maize-Soy supplement)

INTERVENTIONS:
Dietary Supplement: Tenebrio Molitor powder — The intervention consists of a daily dietary supplement made from Tenebrio molito powder, a sustainable and high-protein insect. Each participant in the intervention group will receive a pre-measured daily dose of Tenebrio molitor The supplement is designed to improve protein quality and micronutrient intake, particularly iron, zinc, and vitamin B12, in children aged 2-10 years.
  This intervention differs from traditional nutritional supplements by using Tenebrio molitor as a novel source of animal protein and micronutrients, contributing to sustainable food systems and child nutrition in low-resource settings.
  Arms: Intervention Group
Dietary Supplement: Control Group (Maize-Soy supplement) — The control supplement is a daily dietary mixture made from maize and soy flour, formulated to match the dose of the intervention supplement but without Tenebrio molitor protein. This preparation represents a conventional plant-based dietary supplement commonly used in nutritional support programs.
  It serves as an active comparator to assess the added nutritional and functional benefits of Tenebrio molitor flour in improving biochemical and anthropometric indicators of child nutrition.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to evaluate whether a dietary supplement based on Tenebrio molitor (mealworm flour) can improve nutritional status and biomarkers of micronutrient deficiency in children aged 2-10 years.

The main questions it aims to answer are:

• Does regular supplementation with Tenebrio molitor flour improve chronic malnutrition status

Researchers will compare the intervention group (children receiving Tenebrio molitor flour supplement) with the control group (children receiving a traditional maize-soy flour supplement) to assess differences in biochemical and anthropometric outcomes after the intervention period.

Participants will:

* Participate in baseline and follow-up anthropometric and blood sample assessments (hemoglobin, albumin, zinc, iron, calcium, magnesium, vitamin A, folic acid, vitamin B12, prealbumin).
* Consume a daily dietary supplement (either Tenebrio molitor flour or maize-soy flour) for the duration of the intervention.
* Provide information on dietary intake and general health status through structured questionnaires administered by the research team.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with chronic malnutrition (weight-for-height or BMI below -2 SD according to WHO standards).

Children whose families agree to participate in the intervention and sign the informed consent form.

Exclusion Criteria:

* Children with severe acute illnesses that may interfere with the intervention.
* Children with known allergies to the ingredients of the nutritional products provided.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Prealbumin | Baseline (Week 0) and 24 weeks of supplementation.
  Prealbumin levels will be measured to assess improvement in protein nutritional status among participants receiving Tenebrio molitor flour supplement compared with those receiving maize-soy flour supplement.
Height-for-Age z-scores (WHO Child Growth Standards) | Baseline, 12 weeks and 24 weeks
  To evaluate the effect of Tenebrio molitor supplementation on growth parameters in children. Scale range: z-scores less than or equal to -2 indicate stunting; less than or equal to -3 indicate severe stunting. Values close to 0 reflect adequate growth. High positive values (>+2 or >+3) indicate heights that are significantly above the average

SECONDARY OUTCOMES:
Change in Serum Iron Concentration (µg/dL) | From Baseline to 24 Weeks
  To determine whether Tenebrio molitor flour improves serum iron levels compared to maize-soy flour.
Change in Serum Zinc Concentration (µg/dL) | From Baseline to 24 Weeks
  To determine whether Tenebrio molitor flour improves serum Zinc levels compared to maize-soy flour.
Change in Serum Vitamin B12 Concentration (pg/mL) | From Baseline to 24 Weeks
  To determine whether Tenebrio molitor flour improves serum Vitamin B12 levels compared to maize-soy flour.
Change in Serum Vitamin B9 (Folate) Concentration (µg/dL) | From Baseline to 24 Weeks
  To determine whether Tenebrio molitor flour improves serum Vitamin B9 (Folate) levels compared to maize-soy flour.
Change in Serum Vitamin A Concentration (µg/dL) | From Baseline to 24 Weeks
  To determine whether Tenebrio molitor flour improves serum Vitamin A levels compared to maize-soy flour.
Change in Serum Calcium Concentration (mg/dL) | From Baseline to 24 Weeks
  To determine whether Tenebrio molitor flour improves serum Calcium levels compared to maize-soy flour.
Change in Serum Magnesium Concentration (mg/dL) | From Baseline to 24 Weeks
  To determine whether Tenebrio molitor flour improves serum Magnesium levels compared to maize-soy flour.

CONTACTS AND LOCATIONS:
Overall Officials: Nerea Martín Calvo, Study Director — University of Navarra
Locations (1):
- Kesho Congo, Bukavu, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided